CLINICAL TRIAL: NCT06990581
Title: Effect of Core Exercises on Trunk Stability and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Reem Dawood, Assistant Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Core Stability
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-05

CONDITIONS: Core Stability

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular core group (Experimental): regular core exercises
  Interventions: Other: regular core exercises
- Specific core group (Experimental): specific type of core exercises
  Interventions: Other: specific type of core exercises

INTERVENTIONS:
Other: regular core exercises — regular core exercises on trunk stability and balance
  Arms: Regular core group
Other: specific type of core exercises — specific type of core exercises on trunk stability and balance
  Arms: Specific core group

SUMMARY:
Aim of the study is to investigate the effect of core exercises on trunk stability and balance

DETAILED DESCRIPTION:
participants will be divided into two groups

ELIGIBILITY:
Inclusion Criteria:

* active well-trained female (more than 2 years of training)

Exclusion Criteria:

* any injuries or surgeries in back, lower limbs or upper limbs

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
McGill test | pre and after 6 weeks
Dynamic balance test | pre and after 6 weeks
Maximal strength test | pre and after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Osama R Abdelraouf, PhD, Study Director — Batterjee Medical College
Locations (1):
- Batterjee Medical College, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No